CLINICAL TRIAL: NCT02118675
Title: Tanita® BIA System Validation
Brief Title: Tanita BIA System Validation
Acronym: Tanita
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Tanita (Unknown)
Responsible Party: Principal Investigator, Steven Heymsfield, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 12021
Record Dates: First submitted 2014-04-10; First posted 2014-04-21 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Body Composition; Circumference Measurements; Tissue Thickness Measurements
MeSH Terms: interventions — Body Weights and Measures; Body Composition; Deuterium Oxide; Absorptiometry, Photon; Waist Circumference; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Age 5-17 years: Participants age 5 - 17 will complete the following Body Measurements Body Composition and Circumference Measurements Whole Body DXA Scan Bioelectrical Impedance Analysis (BIA) BodPod Circumferences Ultrasound
  Interventions: Other: Body Measurements; Other: Body Composition and Circumference measurements; Other: Whole Body DXA scan; Other: Bioelectrical Impedance Analysis (BIA); Other: BodPod; Other: Circumferences; Other: Ultrasound
- Age 18-80 years: Participants age 18-80 will complete the following Body Measurements Body Composition and Circumference Measurements Whole Body DXA Scan Bioelectrical Impedance Analysis (BIA) BodPod Circumferences Ultrasound
  Interventions: Other: Body Measurements; Other: Body Composition and Circumference measurements; Other: Whole Body DXA scan; Other: Bioelectrical Impedance Analysis (BIA); Other: BodPod; Other: Circumferences; Other: Ultrasound

INTERVENTIONS:
Other: Body Measurements — A series of body measurements will be taken by trained staff. These measurements include height and weight. These measurements will be completed twice during this time. You will wear a hospital gown and bathing suit for these measurements. Your BMI will be calculated from these measurements.
Other: Body Composition and Circumference measurements — This test is to measure the amount of water in your body. After a fasting urine sample is collected, you will drink a glass of water that has been enriched with an atom called a stable isotope (deuterium). After you drink this non-radioactive heavy water, you will provide urine samples several times over the next 4 hours.
  Other Names: Deuterium Dilution (heavy water)
Other: Whole Body DXA scan — This scan measures the amount of bone, muscle, and fat in your body. The scan will be performed using a whole-body scanner. You will be required to wear a hospital gown, to remove all metal-containing objects from your body, and to lie down on the table. You will be carefully positioned on the table, and your legs will be placed together using two Velcro straps. A scanner emitting low energy X-rays and a detector will pass along your body. You will be asked to remain completely still while the scan is in progress. The scan takes approximately ten minutes.
  Other Names: DXA scan
Other: Bioelectrical Impedance Analysis (BIA) — These tests will measure the amount of fat in your body. You will be asked to change into a hospital gown and to remove all footwear and socks/stockings. Once changed and barefoot, you will be asked to stand on a scale (similar to a large gym scale) and to hold on to hand electrodes on each side of the scale. You will be asked to step off of the scale once the measurement is complete (less than one minute). You will repeat this procedure on three different BIA systems.
Other: BodPod — This test will estimate the amount of fat mass and fat free mass in your body. You will be required to change into a swimsuit and swim cap that we will provide for this procedure. If your swimsuit meets the necessary criteria, you can bring and wear it for the procedure, or PBRC will provide one for you. You will step onto a scale for a quick weight measurement. Next, you will sit inside of the system like you are sitting in a chair. The door of the system will be closed, but you will have a window so that you can see outside of the system while the measurements are completed. The test will be completed in about 15 minutes.
Other: Circumferences — This test will measure the circumferences of your waist, hip, neck, arms, and legs and the lengths of your forearm, upper arm, thigh, and lower leg. The circumference measurements will be made by a trained observer using a calibrated tape measure and an automated circumference measurement device (KX-16). These measurements will be made in about 30 minutes.
  Other Names: KX-16
Other: Ultrasound — An ultrasound is a procedure that uses sound waves to create a picture of an organ or soft tissue. This test measures the size of your tissue thicknesses for fat and skeletal muscle. For this procedure, you will be asked to raise your shirt, disrobe from the waist up, or change into a hospital gown and lie flat on your back on an examination table, or sit on a chair, or stand for measuring your leg dimensions. A gel will be spread on the ultrasound probe, and the probe will be applied directly to the skin on your arms, legs, and abdomen. You will feel slight pressure when the probe is applied. The entire procedure will take approximately 30 minutes.

SUMMARY:
The study is to collect the body composition data using five different methods-bioimpedance analysis (Tanita®), DXA (GE Medical), BodPod (Life Medical), deuterium dilution (heavy water), body circumferences (tape measure, TC2), and tissue thickness by ultrasound (GE Medical, BodyMetrix).

DETAILED DESCRIPTION:
If you are eligible and you choose to participate in this study, you will be asked to come to the Pennington Biomedical Research Center in Baton Rouge between 7:00 and 11:00am after a 10-hour fast (nothing to eat or drink besides water for 10 hours prior to your appointment). The study visit will take approximately five hours. During the visit, you will complete the informed consent process and then complete several body measurements and body composition procedures immediately afterwards.

Description of study procedures

Body Measurements (about 10 minutes):

A series of body measurements will be taken by trained staff. These measurements include height and weight. These measurements will be completed twice during this time. You will wear a hospital gown and bathing suit for these measurements. Your BMI will be calculated from these measurements.

Body Composition and Circumference Measurements Deuterium Dilution (heavy water) This test is to measure the amount of water in your body. After a fasting urine sample is collected, you will drink a glass of water that has been enriched with an atom called a stable isotope (deuterium). After you drink this non-radioactive heavy water, you will provide urine samples several times over the next 4 hours.

Whole Body DXA Scan, about 20 minutes This scan measures the amount of bone, muscle, and fat in your body. The scan will be performed using a whole-body scanner. You will be required to wear a hospital gown, to remove all metal-containing objects from your body, and to lie down on the table. You will be carefully positioned on the table, and your legs will be placed together using two Velcro straps. A scanner emitting low energy X-rays and a detector will pass along your body. You will be asked to remain completely still while the scan is in progress. The scan takes approximately ten minutes.

Bioelectrical Impedance Analysis (BIA) (about 20 minutes):

These tests will measure the amount of fat in your body. You will be asked to change into a hospital gown and to remove all footwear and socks/stockings. Once changed and barefoot, you will be asked to stand on a scale (similar to a large gym scale) and to hold on to hand electrodes on each side of the scale. You will be asked to step off of the scale once the measurement is complete (less than one minute). You will repeat this procedure on three different BIA systems.

BodPod (about 30 minutes) This test will estimate the amount of fat mass and fat free mass in your body. You will be required to change into a swimsuit and swim cap that we will provide for this procedure. If your swimsuit meets the necessary criteria, you can bring and wear it for the procedure, or PBRC will provide one for you. You will step onto a scale for a quick weight measurement. Next, you will sit inside of the system like you are sitting in a chair. The door of the system will be closed, but you will have a window so that you can see outside of the system while the measurements are completed. The test will be completed in about 15 minutes.

Circumferences (about 30 minutes) This test will measure the circumferences of your waist, hip, neck, arms, and legs and the lengths of your forearm, upper arm, thigh, and lower leg. The circumference measurements will be made by a trained observer using a calibrated tape measure and an automated circumference measurement device (KX-16). These measurements will be made in about 30 minutes.

Ultrasound (about 30 minutes) An ultrasound is a procedure that uses sound waves to create a picture of an organ or soft tissue. This test measures the size of your tissue thicknesses for fat and skeletal muscle. For this procedure, you will be asked to raise your shirt, disrobe from the waist up, or change into a hospital gown and lie flat on your back on an examination table, or sit on a chair, or stand for measuring your leg dimensions. A gel will be spread on the ultrasound probe, and the probe will be applied directly to the skin on your arms, legs, and abdomen. You will feel slight pressure when the probe is applied. The entire procedure will take approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Being either male or female
* Being from 5 to 80 years of age
* Being considered normal weight, overweight, or obese based on specified BMI ranges
* Having a bodyweight of less than 440 pounds
* Being willing to comply with the study procedures

Exclusion Criteria:

* Having metal-containing objects in your body
* Being pregnant or attempting to become pregnant
* Being claustrophobic
* Having medical implants such as a pacemaker or metal joint replacements
* Being a professional athlete or someone with severe oedema or dehydration
* Having a body weight greater than 440 pounds

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male or Female age 5 - 80 years of age.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The Primary purpose is to measure children and adult body composition data using different methods - bioimpedance analysis (Tanita®), DXA (GE Medical), BodPod (Life Medical). | One five hour visit (Baseline)
  Tanita® has several Bioelectrical Impedance Analysis (BIA) systems on the market. BIA is considered one of the most reliable and accessible methods of screening body fat. This study will collect data from the Tanita® systems, DXA, BodPod, and total body water to further improve the accuracy of Tanita® products for adults and children.

SECONDARY OUTCOMES:
The secondary outcome measure it to improve the BIA body composition using deuterium dilution (heavy water), body circumferences (tape measure, TC2, Human Solutions), and tissue thickness by ultrasound (GE Medical, BodyMetrix). | One five hour visit (Baseline)
  As part of this analysis additional measurements of body circumferences will be measured with a tape measure and tissue thicknesses by ultrasound will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Heymsfield, MD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States